CLINICAL TRIAL: NCT06447857
Title: Cardiac MRI Extracellular Volume Associated With New-Onset Atrial Fibrillation in Patients With ST-Segment Elevation Myocardial Infarction
Brief Title: Extracellular Volume Associated With New-Onset Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: XYFY2024-KL189-01
Record Dates: First submitted 2024-05-31; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-05

CONDITIONS: Cardiac Magnetic Resonance; Extracellular Volume Overload; Myocardial Infarction; Atrial Fibrillation
MeSH Terms: conditions — Myocardial Infarction; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STEMI underwent CMR: This retrospective study included patients diagnosed with STEMI at the Affiliated Hospital of Xuzhou Medical University.
  Interventions: Other: Cardiac MRI

INTERVENTIONS:
Other: Cardiac MRI — This retrospective study included patients diagnosed with STEMI at the Affiliated Hospital of Xuzhou Medical University. All patients underwent CMR.

SUMMARY:
Left ventricular fibrosis is strongly associated with atrial fibrillation (AF). However, the relationship between LV fibrosis and new-onset AF (NOAF) after ST-segment elevation myocardial infarction (STEMI) is currently unknown. This study was to investigate the relationship between different regions of ECV and NOAF during the acute phase of STEMI. ECV in integral (integral ECV), non-myocardial infarction region (NMI-ECV) and myocardial infarction region (MI-ECV) was obtained by CMR.

DETAILED DESCRIPTION:
This retrospective study included patients diagnosed with STEMI at the Affiliated Hospital of Xuzhou Medical University. All patients underwent CMR during hospitalization, which included T1 mapping sequences. The blood sampling was collected within 24 hours of the CMR examination. Inclusion criteria: 1. Successful pPCI (TIMI flow ≥ 2) within 12 hours after symptom onset; 2. Admission to the cardiac care unit for continuous electrocardiogram (ECG) monitoring after pPCI. Exclusion criteria: 1. Poor image quality; 2. History of myocardial infarction; 3. History of atrial fibrillation; 4. Malignancy, or inflammatory disease; 5. Severe valvular heart disease; 6. Thyroid dysfunction. NOAF was defined as post-admission atrial fibrillation without a history of atrial fibrillation. ECG monitoring revealed a suspicious rhythm during admission, and an immediate 12-lead ECG confirmed NOAF. Infarct-related arteries (IRA) were recorded based on CAG findings. ECV in integral (integral ECV), non-myocardial infarction region (NMI-ECV) and myocardial infarction region (MI-ECV) was obtained by CMR.

ELIGIBILITY:
Inclusion Criteria:

* Successful pPCI (TIMI flow ≥ 2) within 12 hours after symptom onset
* Admission to the cardiac care unit for continuous electrocardiogram (ECG) monitoring after pPCI

Exclusion Criteria:

* Poor image quality
* History of myocardial infarction
* History of atrial fibrillation
* Malignancy, or inflammatory disease
* Severe valvular heart disease
* Thyroid dysfunction

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective study included patients diagnosed with STEMI at the Affiliated Hospital of Xuzhou Medical University from January 2020 to May 2024. All patients underwent CMR during hospitalization, which included T1 mapping sequences. The blood sampling was collected within 24 hours of the CMR examination. NOAF was defined as post-admission atrial fibrillation without a history of atrial fibrillation. ECV in integral (integral ECV), non-myocardial infarction region (NMI-ECV) and myocardial infarction region (MI-ECV) was obtained by CMR.
Sampling Method: Non-Probability Sample
Enrollment: 589 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Primary endpoint events included new-onset atrial fibrillation | during hospitalization (assessed up to 10 days)
  NOAF was defined as post-admission atrial fibrillation without a history of atrial fibrillation. ECG monitoring revealed a suspicious rhythm during admission, and an immediate 12-lead ECG confirmed NOAF.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No